CLINICAL TRIAL: NCT00525486
Title: Extended Release Nifedipine Treatment as Maintenance Tocolysis to Prevent Preterm Delivery:A Prospective Interventional Study
Brief Title: Extended Release Nifedipine Treatment as Maintenance Tocolysis to Prevent Preterm Delivery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: The Baruch Padeh Medical Center, Poriya (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PTL prevention Nifedipine
Record Dates: First submitted 2007-09-02; First posted 2007-09-05 (Estimated); Last update posted 2010-12-23 (Estimated); Status verified 2010-12

CONDITIONS: Preterm Labor
Keywords: Nifedipine; Tocolysis; Maintenance; Preterm delivery; extended release nifedipine; PTL
MeSH Terms: conditions — Obstetric Labor, Premature; Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): The treated group of pregnant women, after having successful treatment for PTL
  Interventions: Drug: Nifedipine extended release
- B (No Intervention): The no treatment arm of women treated with tocolysis for PTL.

INTERVENTIONS:
Drug: Nifedipine extended release — Nifedipine extended release PO 30 mg X2/d until 34 weeks' gestation
  Other Names: Osmo-Adalat 30 mg
  Arms: A

SUMMARY:
To evaluate the treatment efficacy and safety usig extended release nifedipine, as maintenance therapy to pregnant women who were hospitalized and treated for preterm labor until 34 weeks' gestation. After the PTL will stop, we will randomize these women for the treatment group and the control (no treatment) group.

The main outcome will be preterm delivery before 34 weeks' gestation. the secondary outcome will be the side effects of the medication and the newborn/mother health variables.

ELIGIBILITY:
Inclusion Criteria:

* pregnancy week 24-33
* Singleton pregnancy
* After successful treatment to stop PTL

Exclusion Criteria:

* Contraindications for Nifedipine extended release treatment.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2007-12

CONTACTS AND LOCATIONS:
Overall Officials: Yuri Perlitz, MD, Principal Investigator — The Baruch Padeh Medical Center, Poria, Israel.

REFERENCES:
- [Derived] Wilson A, Hodgetts-Morton VA, Marson EJ, Markland AD, Larkai E, Papadopoulou A, Coomarasamy A, Tobias A, Chou D, Oladapo OT, Price MJ, Morris K, Gallos ID. Tocolytics for delaying preterm birth: a network meta-analysis (0924). Cochrane Database Syst Rev. 2022 Aug 10;8(8):CD014978. doi: 10.1002/14651858.CD014978.pub2. PMID 35947046